CLINICAL TRIAL: NCT07387523
Title: Psychological and Lifestyle Factors That Predict Adherence of Multi-domain Interventions for Promoting Brain Health
Acronym: ToBrainHealth
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gabriele Cattaneo (Other)
Collaborators: Universidad Politecnica de Madrid (Other)
Responsible Party: Sponsor-Investigator, Gabriele Cattaneo, PhD, Institut Guttmann
Organization: Institut Guttmann (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CEI 25/46; PID2022-139298OA-C22 (Other Grant/Funding Number: Spanish Ministry of Science and Innovation)
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Brain Health; Cognition; Healthy Adult Participants
Keywords: brain health, adherence, intervention, mHealth, lifestyles

STUDY DESIGN:
Intervention Model Description: The study uses a three-arm, parallel-group interventional design in which 120 participants from the Barcelona Brain Health Initiative cohort are pseudo-randomly allocated (stratified by age and sex) to one of three conditions: (1) a control group receiving generic, non-personalized lifestyle education; (2) a personalized digital intervention delivered through the ToBrainHealth platform; or (3) a personalized digital intervention plus intensive professional coaching. All groups participate concurrently over an 8-week period. The design allows comparison of increasing levels of personalization and support to determine their relative effectiveness in improving adherence to healthy lifestyle behaviors and in producing changes in clinical, cognitive, and psychosocial outcomes.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants remain blinded to their intervention assignment. Group allocation is determined by the principal investigator and kept in sealed envelopes. At the baseline visit, the evaluator opens the envelope immediately before administering the assessments; therefore, evaluators are not blinded during the assessment itself but remain unaware of the assignment until that moment. Other study personnel not involved in delivering the intervention (e.g., data analysts) remain masked throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Generic Lifestyle Education (Sham Comparator): Participants receive general, non-personalised educational materials about healthy lifestyle habits, including information on nutrition, physical activity, sleep, cognitive stimulation and psychological wellbeing. They do not receive personalised recommendations nor access to adaptive features of the ToBrainHealth platform. Participants complete periodic online questionnaires to report their activities, but no tailored guidance or coaching is provided.
  Interventions: Behavioral: Generic Lifestyle Education
- Digital Personalised Intervention (Active Comparator): Participants use the ToBrainHealth digital platform, which provides personalised lifestyle recommendations based on individual behavioural and psychological profiles. The platform delivers adaptive intervention strategies, remote asynchronous monitoring and feedback. Participants also wear a Fitbit HR device that synchronises activity and sleep data with the platform. No human coaching is provided; all support is delivered digitally through the platform's personalised features.
  Interventions: Behavioral: ToBrainHealth Personalised Digital Intervention
- Digital Personalised Intervention + Coaching (Experimental): Participants receive the full personalised digital intervention described for Arm 2, including tailored recommendations, adaptive strategies, digital monitoring and wearable integration. In addition, they receive intensive professional health coaching throughout the 8-week programme. Coaching sessions aim to enhance motivation, address barriers to behaviour change, reinforce adherence and optimise long-term adoption of healthy lifestyle habits.
  Interventions: Behavioral: ToBrainHealth Personalised Digital Intervention with Coaching

INTERVENTIONS:
Behavioral: Generic Lifestyle Education — Participants receive non-personalized educational materials about healthy lifestyle habits related to brain health. They complete periodic questionnaires but do not receive individualized recommendations, adaptive digital support, or coaching. This condition serves as a comparison group to evaluate the added benefit of personalized digital interventions.
  Arms: Generic Lifestyle Education
Behavioral: ToBrainHealth Personalised Digital Intervention — This intervention uses the ToBrainHealth digital platform to deliver personalised lifestyle recommendations and adaptive behaviour-change strategies based on each participant's psychological and behavioural profile. The platform integrates data from a Fitbit HR wearable to monitor activity and sleep. Guidance and monitoring are entirely digital, with no human coaching provided.
  Arms: Digital Personalised Intervention
Behavioral: ToBrainHealth Personalised Digital Intervention with Coaching — This intervention includes the full personalised digital program described above, enhanced with intensive, structured health coaching delivered by trained professionals. Coaching sessions aim to support motivation, address individual barriers, and reinforce adherence to lifestyle recommendations. This arm allows assessment of the added value of professional guidance beyond digital personalisation alone.
  Arms: Digital Personalised Intervention + Coaching

SUMMARY:
Ageing is associated with a rising burden of neurological disorders, particularly dementia, which are now the leading cause of disability worldwide. Many dementia cases could potentially be prevented by modifying lifestyle factors such as physical inactivity, unhealthy diet, poor sleep, low social engagement and psychological distress. The Barcelona Brain Health Initiative (BBHI), a longitudinal cohort of more than 6,000 adults aged 40-75 years, has shown substantial inter-individual variability in lifestyle and psychological profiles and has identified subgroups at higher risk for poorer brain health.

ToBrainHealth is an 8-week, three-arm controlled intervention nested within BBHI. It evaluates different levels of personalisation and support to optimise healthy lifestyle behaviours using the ToBrainHealth platform, a digital platform that delivers recommendations, collects self-reported behaviours and integrates data from wearable activity trackers.

A total of 120 BBHI volunteers classified as moderate- or high-risk based on previous lifestyle and psychological questionnaires will be selected (40 per arm). Allocation to study arms will be pseudo-randomised, stratified by age, sex, and lifestyle and psychological profiles.

The three groups are: (1) a control group receiving only generic, non-personalised education about healthy lifestyles and regular online questionnaires, without use of ToBrainHealth platform tailoring; (2) a digital personalised intervention group using ToBrainHealth platform to deliver tailored lifestyle recommendations, adaptive intervention strategies and remote asynchronous supervision, supported by data from questionnaires and wearables; and (3) a digital personalised intervention plus intensive health-coaching group, which receives the same ToBrainHealth platform-based programme plus structured, proactive support and supervision by health professionals to enhance motivation and adherence.

The primary outcome is adherence to the lifestyle intervention, operationalised as the percentage of recommended activities and goals achieved during the 8-week programme, based on platform's logs, questionnaires and wearable data. The study will test whether lifestyle and psychological profile increases adherence compared with generic education, and whether adding intensive coaching provides additional benefit (expected gradient: coaching > digital only > control).

Secondary outcomes include the clinical impact of the intervention on brain-health-related measures. All participants will undergo pre- and post-intervention assessments including a brief medical evaluation (vital signs and anthropometrics), a digital neuropsychological battery, and questionnaires on motivation, lifestyle and psychosocial variables. These data will be analysed together with existing BBHI longitudinal information to explore changes in cognitive performance, health status and psychological wellbeing, and to characterise patterns and predictors of adherence across intervention arms.

The trial will also assess feasibility and acceptability of ToBrainHealth platform as a remote monitoring and coaching tool for brain-health promotion. Results are expected to generate new knowledge on the role of psychological and lifestyle profiles in adherence, and to inform scalable, technology-supported, personalised interventions aimed at preserving brain health and reducing the long-term risk of cognitive decline in community-dwelling adults.

DETAILED DESCRIPTION:
ToBrainHealth Intervention Trial - Three-arm personalised lifestyle optimisation study The ToBrainHealth intervention trial is an 8-week, three-arm controlled study designed to evaluate the impact of personalised, technology-supported strategies on adherence to healthy lifestyle recommendations in community-dwelling adults. The study is embedded in the Barcelona Brain Health Initiative (BBHI), a large longitudinal cohort that investigates determinants of brain health across ageing. The trial addresses a crucial challenge in brain-health promotion: despite strong evidence that modifiable lifestyle factors positively influence resilience and reduce the risk of cognitive decline, long-term adherence to lifestyle interventions remains low.

Background and Rationale Ageing is associated with increasing prevalence of neurological disorders, particularly dementia, which represent the leading cause of disability globally. Cognitive decline is not inevitable; ~20% of older adults maintain youthful cognitive performance, reflecting brain resilience processes. Research from the BBHI cohort (>6,000 adults aged 40-75 years) demonstrates that lifestyle quality, psychological wellbeing, sleep, social engagement and physical activity predict brain health trajectories. However, substantial variability exists between individuals.

To better understand this variability, latent profile analysis of lifestyle and psychosocial data from the BBHI cohort identified three behavioural-psychological profiles: High Risk, Moderate Risk and Low Risk. High- and Moderate-Risk individuals exhibit poorer habits and lower levels of protective traits such as sense of coherence, self-reflection or emotional wellbeing, all of which influence adherence. These profiles provide an empirical basis for targeted interventions.

Lifestyle interventions often fail due to barriers such as lack of personalisation, limited feedback, insufficient motivational support, technical difficulties, and fluctuating emotional states. Evidence shows that technology-supported programmes can enhance adherence when they provide clear guidance, personalised content, adaptive strategies, monitoring features, and-when appropriate-professional supervision. The ToBrainHealth digital solution operationalises this knowledge to deliver multimodal lifestyle recommendations tailored to each participant's psychological and behavioural profile.

Study Objectives

Primary objective:

To determine whether digital personalisation and professional coaching improve adherence to a lifestyle-optimisation intervention.

Secondary objectives:

1. Evaluate whether personalisation delivered through the ToBrainHealth platform increases adherence compared to generic, non-personalised education.
2. Assess the added value of intensive health coaching when combined with a personalised digital intervention.
3. Measure clinical impact via pre- and post-intervention medical, neuropsychological and psychosocial assessments.
4. Assess feasibility and acceptability of the ToBrainHealth platform as a remote monitoring and intervention tool.
5. Analyse adherence patterns and identify demographic, psychological and motivational factors influencing response to different intervention intensities.

Study Design This is a controlled, three-arm intervention trial lasting 8 weeks. A total of 120 participants will be selected from the BBHI cohort among those classified into the High-Risk and Moderate-Risk latent profiles based on recent lifestyle, personality, and psychological questionnaires. Sixty individuals from each risk profile will be randomly selected. They will then be pseudo-randomised, stratified by age and biological sex, and psychological profile into one of the three study arms (n=40 per arm). Allocation will be concealed until the first visit, where each participant receives the appropriate study documentation.

Intervention Arms

1. Control group - Generic lifestyle education (no technology) Participants receive non-personalised educational materials on healthy lifestyle habits. They periodically complete online questionnaires but do not receive any personalised recommendations or digital-driven adaptive strategies.
2. Personalised Digital Intervention - ToBrainHealth platform (no personal coach)

   Participants use the ToBrainHealth platform, a technology-based solution developed by Institut Guttmann and the Universidad Politécnica de Madrid, which allows:
   * Personalised lifestyle recommendations based on behavioural and psychological profiles.
   * Adaptive intervention strategies that evolve according to user engagement and progress.
   * Remote, asynchronous monitoring of behavioural changes.
   * Integration of multimodal lifestyle information (cognitive activities, nutrition, sleep, socialisation, psychological state, physical activity).

   Participants also wear a Fitbit HR device, synchronised with the platform to collect activity and sleep metrics. The device is loaned exclusively for study participation and must be returned upon completion.
3. Personalised Digital Intervention + Intensive Coaching - ToBrainHealth platform This arm receives exactly the same personalised digital intervention described in Arm 2, complemented by intensive professional health coaching. Coaching aims to enhance motivation, address barriers to engagement, reinforce adherence, and support the adoption of long-lasting healthy behaviours.

Outcome Measures Primary Outcome: Adherence

Adherence is quantified as the percentage of recommended lifestyle actions completed during the 8-week intervention. The study will evaluate:

* Whether personalised digital guidance enhances adherence compared to the generic control group.
* Whether intensive coaching produces additional improvements beyond digital personalisation alone.

Secondary Outcomes: Clinical Impact and Behavioural Change

Before and after the 8-week intervention, all participants undergo standardised assessments, including:

Medical evaluation

* General health status, anthropometry (weight, height) and blood pressure. Neuropsychological evaluation
* Computer-based tasks measuring attention, memory, processing speed and executive function.

Motivational and lifestyle assessment

- Used to refine personalised recommendations and characterise motivational profiles.

Results from these evaluations will be integrated with the extensive longitudinal information already available from the BBHI cohort, allowing analysis of changes in cognitive performance, psychological wellbeing and lifestyle patterns.

Sample Size and Statistical Considerations The total sample size (n=120) reflects power calculations based on expected small-to-moderate intervention effects (d≈0.3) observed in previous coaching-based lifestyle studies. With α=0.05 and power of 80%, the required sample is ~110 participants; 120 are recruited to compensate for an estimated 10% attrition rate. Planned analyses include repeated-measures ANOVAs and general linear models to compare intervention effects within and between groups.

Data Management and Confidentiality All data will be managed using dedicated REDCap electronic case-report forms. Data will be pseudonymised using unique participant codes. Identifiable information will be stored separately with restricted access and password-protected systems. Audit trails will document all modifications. Data export for statistical analysis will follow controlled procedures and comply with GDPR (Regulation EU 2016/679) and Spanish data-protection legislation (LO 3/2018). Fitbit data synchronisation requires explicit participant authorisation.

Regular data backups and REDCap system audits are performed at Institut Guttmann to guarantee data integrity and security.

Ethical Considerations Participants receive detailed written and verbal information about the study, including procedures, duration, potential risks, benefits, and data-protection safeguards. Participation is voluntary, and withdrawal may occur at any moment without explanation or consequences. No participant can be included without providing signed informed consent. The study protocol is submitted to the corresponding Research Ethics Committee (CER) prior to initiation, and any non-administrative protocol amendments require CER approval.

Implementation Schedule

The project includes:

* Parallel implementation of the three intervention arms, including baseline assessments, 8-week intervention period and follow-up evaluations.
* Data analysis and preparation of scientific publications.

Expected Scientific and Societal Impact The ToBrainHealth digital solution aims to advance understanding of resilience mechanisms and behaviour-change processes relevant to brain health. By combining personalisation, remote monitoring, digital phenotyping and intensive coaching, the study aspires to produce evidence-based, scalable strategies for maintaining brain health across the lifespan. Findings are expected to inform the development of personalised preventive programmes and guide public-health approaches aimed at reducing long-term risk of cognitive decline in ageing populations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult participating in the Barcelona Brain Health Initiative

Exclusion Criteria:

* Neurological or psychiatric disease

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to Recommended Healthy Lifestyle Activities | From baseline to the end of the 8-week intervention period.
  Adherence will be defined as the percentage of recommended healthy lifestyle activities (e.g., physical activity, cognitive training, sleep routines, social and psychological exercises) that each participant completes during the 8-week intervention. It will be calculated from ToBrainHealth platform logs, self-reported questionnaires and Fitbit HR data, summarised as an overall adherence score for each participant and compared across intervention arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Guttmann Barcelona. Institut de Salut Cerebral i Neurorehabilitació, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly at this stage. The dataset contains sensitive health and neuropsychological information, and full anonymization without risk of re-identification cannot be guaranteed. In addition, participant consent does not currently include provisions for broad data sharing. Aggregated results will be made publicly available through publications and reports. Future data sharing with qualified researchers may be considered upon reasonable request, subject to ethical approval, data protection regulations, and appropriate data-use agreements.